CLINICAL TRIAL: NCT00765934
Title: Does Rapydan Influence Routine Clinical Chemistry and Hematology Measurements?
Brief Title: Influence of Rapydan on Clinical Chemistry and Hematology Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LabNoord (Other)
Responsible Party: R.F.M. Oude Elferink, LabNoord
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RapydanClinicalChemistry
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Healthy
Keywords: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rapydan (Other): Internal control. Blood from both arms will be drawn. Only one arm of the subject is treated with Rapydan.
  Interventions: Drug: Rapydan

INTERVENTIONS:
Drug: Rapydan — lidocaine / tetracaine 70/70 mg patch
  Other Names: Lidocaine Tetracaine Patch

SUMMARY:
There is an increasing awareness of the importance of treating procedure-related pain. Patients undergoing vascular access procedures are often afraid of needles and the discomfort associated with injections. This type of pain and/or fear can be stressful to patients. [1] For prevention of the pain associated with these procedures, the hospital is using Rapydan plasters. Rapydan consists out of two local anesthetics: lidocaine and tetracaïne. Rapydan produces topical anesthesia after an application time of 30 minutes and is used in the Martini Hospital for pain relieve by venipuncture and IV cannulation. The venous blood draining the anaesthetized skin contains a higher blood concentration of the local anesthetics than does venous blood in other parts of the body [2] Although the concentrations of the local anesthetics are low in patients with normal skin, the question is whether the presence of the local anesthetics which Rapydan contains might influence routine measurements in clinical chemistry and hematology.

ELIGIBILITY:
Inclusion Criteria:

Volunteers 20-60 years who are decision making competent

Exclusion Criteria:

Patients with local anesthetic allergy Patients using antiarrhythmic drugs Patients using other local anesthetics

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Routine Clinical Chemistry measurements differences | 1

CONTACTS AND LOCATIONS:
Overall Officials: Rob Oude Elferink, MSc, Study Director — LabNoord
Locations (1):
- LabNoord, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Background] Curry SE, Finkel JC. Use of the Synera patch for local anesthesia before vascular access procedures: a randomized, double-blind, placebo-controlled study. Pain Med. 2007 Sep;8(6):497-502. doi: 10.1111/j.1526-4637.2006.00204.x. PMID 17716323
- [Background] Amdisen A, Glud V. No influence from topical application of EMLA cream before blood sampling on routine clinical chemistry and haematology measurements. Eur J Clin Pharmacol. 1991;41(6):619-20. doi: 10.1007/BF00314997. PMID 1815978